CLINICAL TRIAL: NCT00870532
Title: A Prospective Study of Metronomic Oral Vinorelbine in Combination With Sorafenib in Advanced Non-small Cell Lung Cancer a) A Phase I Dose-finding Study of the Combination of Metronomic Oral Vinorelbine and Sorafenib b) Pharmacokinetics Profiling of the Combination of Metronomic Oral Vinorelbine and Sorafenib at MTD
Brief Title: Study of Combination of Metronomic Oral Vinorelbine and Sorafenib in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Eng-Huat Tan, Senior Consultant, National Cancer Centre, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-3-LUN
Record Dates: First submitted 2008-06-09; First posted 2009-03-27 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Phase I; Combination; Anti-angiogenic; Sorafenib; Metronomic oral vinorelbine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 60 mg/week of vinorelbine + sorafenib
  Interventions: Drug: oral vinorelbine; Drug: sorafenib
- 2 (Experimental): 90 mg/week of vinorelbine + sorafenib
  Interventions: Drug: oral vinorelbine; Drug: sorafenib
- 3 (Experimental): 120 mg/week of vinorelbine + sorafenib
  Interventions: Drug: oral vinorelbine; Drug: sorafenib

INTERVENTIONS:
Drug: oral vinorelbine — The patients will be divided into 3 cohorts (15 patients per cohort), each cohort receiving a fixed metronomic (thrice a week) dose of oral vinorelbine at 60 mg/week, 90 mg/week, and 120 mg/week respectively. We should arrive at 3 different MTDs from the 3 cohorts.
  Other Names: Navelbine Oral
Drug: sorafenib — Each patient within each cohort will receive a starting dose of sorafenib at 200 mg bid for 4 weeks. In the absence of dose-limiting toxicities, the dose of sorafenib will be escalated to 400 mg bid for another 4 weeks, 600 mg bid for 4 weeks and then finally 800 mg bid. We should arrive at 3 different MTDs from the 3 cohorts.
  Other Names: Nexavar

SUMMARY:
Targeting the blood supply of cancer, called anti-angiogenesis is a new but proven treatment strategy. There are two ways of achieving this effect. The first way to specifically target the molecular pathways that promote new blood vessel formation in cancer. An example of such an agent is sorafenib, which is an oral agent and which is already in use worldwide for the treatment of kidney and liver cancers. The second way is to target the cells lining the blood vessels by using low dose of chemotherapy agents administered at frequent intervals. This strategy is called metronomic chemotherapy. It is possible that combining agents like sorafenib and metronomic chemotherapy may further enhance anti-cancer effects. This study aims to determine the optimal way of combining oral vinorelbine in metronomic doses and sorafenib. Oral vinorelbine is a chemotherapy agent that is already approved for use in cancer treatment such as lung cancer. By combining both oral anti-cancer agents to optimize their anti-angiogenic effects in this study, the potential benefit to the patients can be tremendous and far-reaching. Special radiologic imagings and blood tests will be incorporated into this study to help further the understanding of the anti-angiogenic processes of both agents.

DETAILED DESCRIPTION:
Phase I Dose-finding study: The patients will be divided into 3 cohorts (15 patients per cohort), each cohort receiving a fixed metronomic (thrice a week) dose of oral vinorelbine at 60 mg/week, 90 mg/week, and 120 mg/week respectively. Each patient within each cohort will receive a starting dose of sorafenib at 200 mg bid for 4 weeks. In the absence of dose-limiting toxicities, the dose of sorafenib will be escalated to 400 mg bid for another 4 weeks, 600 mg bid for 4 weeks and then finally 800 mg bid. We should arrive at 3 different MTDs from the 3 cohorts.

Once the MTD has been determined for each cohort, we will recruit an additional 12 patients for each cohort and study the PK profile of both drugs. The 12 patients in each cohort will be sequentially alternated to group 1 or group 2 treatment schedules. Group 1 (N=6 patients in each cohort) will receive vinorelbine three times per week starting on Monday (Day 1) followed by Wednesday (Day 3) and Friday (Day 5). In the subsequent weeks vinorelbine will be given on the same working days (i.e. Monday, Wednesday and Friday). The first PK profile of vinorelbine (without concomitant sorafenib) will be determined on Day 15 under steady state conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed NSCLC
2. At least one or 2 prior lines of chemotherapy, including oral EGFR tyrosine-kinase inhibitor for metastatic disease or locally advanced unresectable disease. There should be at least 4 weeks since prior chemotherapy or radiation therapy; patients who decline conventional chemotherapy or oral EGFR tyrosine-kinase inhibitor as salvage 2nd or 3rd line treatment are also eligible.
3. Minimum body-surface area (BSA) of 1.4 m2 at point of recruitment. This is a safeguard against recruiting small-built patients who may experience adverse reaction on absolute dosing of oral vinorelbine. At this body surface area, the maximum dosing of oral vinorelbine at 120 mg/week is equivalent to 86 mg/m2/week for a patient with BSA of 1.4 m2.
4. Age >21 years
5. ECOG performance status <2 (Karnofsky >60%)
6. Patients must have normal organ and marrow function as defined here: leukocytes >3,000/mcL, absolute neutrophil count >1,500/mcL, platelet count > 100,000/mcL, serum bilirubin within normal institutional limits, AST(SGOT)/ALT(SGPT) <2.5 X upper limit of normal, and creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients. These tests must be done within 1 week of study treatment.
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
2. Patients receiving any other investigational agents
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Oral Vinorelbine or other agents used in study
5. Prior and / or concomitant treatment with drugs known to induce or inhibit cytochrome P450 3A4: phenytoin, carbamazepine, barbiturates, rifampicin, imidazole antifungals (such as ketoconazole, fluconazole, itraconazole, metronidazole), omeprazole and ritonavir. Patients who are taking gastric acid-lowering agents such as H2 antagonist or antacids will be evaluated regarding the need to continue with these medications. If discontinuation of these medications is medically contraindicated, the patient will be excluded as these agents are known to lower the solubility of sorafenib and hence may limit their efficacy.
6. Significant malabsorption syndrome or disease affecting the gastro-intestinal tract function
7. Significant peripheral or autonomic neuropathy affecting sensation or bowel motility
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
9. Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg despite optimal management
10. Pregnancy or breast-feeding or women of childbearing potential not using effective contraception
11. Evidence or history of bleeding diathesis or coagulopathy
12. Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months
13. Pulmonary hemorrhage/bleeding event >CTCAE grade 2 within 4 weeks of recruitment
14. Any other hemorrhage/bleeding event >CTCAE grade 3 within 4 weeks of recruitment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-06; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
to determine the optimal combination of metronomic oral vinorelbine with sorafenib to achieve anti-angiogenic and hence anti-tumour effect in patients with advanced NSCLC | every 1-2 monthly with DCE-MR and circulating endothelial cells apart from routine CT scans

SECONDARY OUTCOMES:
To determine the response rate to the combination of metronomic oral vinorelbine and sorafenib in advanced NSCLC | CT scan every 2 months while on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eng-Huat Tan, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore